CLINICAL TRIAL: NCT07213440
Title: Identification of Early Markers for ALS
Acronym: PremodiALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C23-41; IDRCB (Registry Identifier: 2024-A00273-44)
Record Dates: First submitted 2025-01-08; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Spinal Puncture; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: 3 groups will be recruited in this study: a pre-symptomatic patient with a genetic mutation responsible for ALS, a control group and a final group of patients with precose ALS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- a single arm (Other): all 3 patient groups will have the same tests
  Interventions: Procedure: lumbar puncture

INTERVENTIONS:
Procedure: lumbar puncture — After information and consent by the investigator, clinical data will be collected using a CRF and biological samples (Blood sampling, Urine sample, cephalo spinal fluid), lacrimal fluid sampling, and a smell test will be taken from all subjects at baseline and at 12 months.
  Other Names: Blood sampling,Urine sample,survey,Lacrimal fluid sampling,Smell test

SUMMARY:
Although several molecules have been proposed as biomarker candidates, a clinically established signature for an early or even premotor diagnosis of ALS is not available. Due to the already advanced, disease stage at the time of diagnosis as well as rapid disease progression, an early diagnosis is mandatory for efficacious disease-modifying therapies.

In this project, the investigators will develop a clinical molecular fingerprint of PGMC that will provide insight into the molecular pathogenesis of ALS and allow earlier diagnosis.

ELIGIBILITY:
Inclusion Criteria:

FIRST GROUP: Premotor gene mutation carriers (PGMC):

* 18-90 years of age
* Provision of a written informed consent
* Affiliation with a social security scheme or beneficiary of such a scheme
* Diagnosed by a clinically certified laboratory with a disease- causing mutation in a known ALS gene by predictive genetic testing
* No symptoms of motor neuron disease explainable otherwise than by mutation in a known ALS gene

SECOND GROUP: Control subjects to premotor gene mutation carriers (CTR):

* 18-90 years of age
* Provision of a written informed consent
* Affiliation with a social security scheme or beneficiary of such a scheme
* No known genetic mutation and no known ALS disease in close family
* No diagnosed motor-neuron disease

THIRD GROUP: ALS (EALS) / ALS mimics (MIM)

* 18-90 years of age
* provision of a written informed consent
* affiliation with a social security scheme or beneficiary of such a scheme
* Patients with pure motor symptom or early ALS (EALS) or ALS mimics (MIM)

EALS are patients with pure motor symptom / early motor symptoms of ALS, including those, where the diagnosis of ALS can already be made. These may be patients who meet the following criteria:

According to El Escorial criteria : patients who can be classified as possible ALS or those who show upper motor neuron (UMN) signs only or lower motor neuron (LMN) signs only, so that classification as possible ALS is also not possible. Symptoms should not persist for more than 12 months.

According to Gold Coast criteria: Patients who do not fulfill the criterion of temporal progression or patients who only show UMN signs or only LMN signs in one region and thus do not fulfill the diagnostic criteria of ALS.

Exclusion Criteria:

* Inability to express consent to the study
* Persons subject to a judicial safeguard measure, under guardianship or curatorship.
* Linguistic incapacity or psychic refusal to read the information.
* Pregnant women
* Foreseen inability to attend scheduled visits
* Persons refusing to take one of the following samples: Acquisition of blood samples, Acquisition of tear fluid samples, Acquisition of urine sample

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Differential proteome from plasma, tear fluid, Cerebrospinal fluid | Baseline, 1 year
  Proteome (DIA-MS) from plasma, tear fluid and cerebrospinal fluid in Premotor gene mutation carriers vs. Control group and Early ALS vs. ALS Mimics
Differential metabolome from plasma, urine , Cerebrospinal fluid | Baseline, 1 year
  Metabolome (LC-MS/MS) from plasma, Urine and cerebrospinal fluid in Premotor gene mutation carriers vs. Control group and Early ALS vs. ALS Mimics
Nf-L, tau/phospho-tau, GFAP (SIMOA) from plasma and CSF | Baseline, 1 year
  Nf-L (Neurofilament light protein), tau/phospho-tau, GFAP from plasma and CSF in Premotor gene mutation carriers vs. Control group and Early ALS vs. ALS Mimics. By SIMOA technology
Soluble p75ECD (ELISA) from urine | Baseline, 1 year
  Soluble p75ECD (ELISA) from urine in Premotor gene mutation carriers vs. Control group and Early ALS vs. ALS Mimics.
B-SIT score (0-12 pts.) | Baseline, 1 year
  Brief Smell Identification Test B-SIT score (0-12 pts.) in Premotor gene mutation carriers vs. Control group and Early ALS vs. ALS Mimics.
Questionnaire | Baseline, 1 year
  Complete a Questionnaire with health data In Premotor gene mutation carriers vs. Control group and Early ALS vs. ALS Mimics.
ECAS-score | Baseline, 1 year
  Cognitive assesment Edinburgh Cognitive and Behavioural ALS Screen-score In Premotor gene mutation carriers vs. Control group and Early ALS vs. ALS Mimics.
Standardized neurological examination by ALSFRS-R (Revised Amyotrophic Lateral Sclerosis Functional Rating Scale) | Baseline, 1 year
  ALSFRS is an instrument for evaluating the functional status of patients with Amyotrophic Lateral Sclerosis.Neurological. Assessment in Premotor gene mutation carriers vs. Control group and Early ALS vs. ALS Mimics. Minimum score 0, maximum score 40
Standardized neurological examination by Manual Muscle Testing (MMT) | Baseline, 1 year
  Manual Muscle Testing provides helpful information about muscle quality. Grade 0 : no concentration palpable to Grade 5 : normal strength.
  Assessment in Premotor gene mutation carriers vs. Control group and Early ALS vs. ALS Mimics.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Tours, Tours, France, France

IPD SHARING:
Plan to Share IPD: No